CLINICAL TRIAL: NCT03215238
Title: Intraoperative Pleth Variability Index (PVI) Variability
Status: Terminated | Type: Observational
Why Stopped: enrollment too slow
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PT1701
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Intraoperative Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- neurosurgical patients: Neurosurgical patients undergoing craniotomies for tumor. 25 subjects
- Neurointerventional patients: Patients undergoing neurointerventional procedures under general anesthesia. 25 subjects

SUMMARY:
Pleth Variability Index (PVI) is a variable that is derived from photoplethysmography (PPG) signal. It is used as a surrogate for intravascular volume status intraoperatively. PVI can have significant amount of baseline variability which appears to oscillate at a very low frequency (5-10 minute cycles). This study aims to investigate the origin of these baseline oscillations.

DETAILED DESCRIPTION:
PVI is derived from the infrared photoplethysmography signal. Intraoperatively during mechanical ventilation it reflect fluid responsiveness which is a surrogate endpoint of intravascular volume.

PVI signal appears to have significant baseline variability which can not be explained by rapid changes in intravascular fluid volume. The baseline PVI changes also appear to oscillate at a very low frequency, much below any previously identified spontaneous vascular oscillations.

The aim of this study is to investigate weather the PVI variability originates from changes in the infrared photoplethysmography signal or if they are possibly due to the algorithm calculating PVI.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical patients for tumor resection
* neurointerventional patients
* general anesthesia with mechanical ventilation
* communicates in english (consent)
* over 18 years of age

Exclusion Criteria:

* unable to sign consent
* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical and neurointerventional patients will be enrolled as these patients do rarely have sudden intravascular volume changes. Neurointerventional patients typically have no significant intravascular fluid changes, but do not routinely have intra-arterial catheters. Neurosurgical patients have slow, steady fluid shifts due to mannitol administration. Since most all of these patients have intra-arterial cannulas, it allows arterial waveform data collection which can be compared to the PPG signal.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
PVI variability | 1 hour
  PVI variability will be compare to raw infrared photoplethysmography signal

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Talke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No